CLINICAL TRIAL: NCT05699512
Title: What is the Prognosis of Functional Ability, Symptoms and Quality of Life in Patients That Are Treated in a University Hospital Because Symptoms of Post Covid-19 Condition
Brief Title: Functional Ability, Symptoms and Quality of Life in Patients With Post Covid-19 Condition
Acronym: LC-cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Helena Liira, Chief Physician, Helsinki University Central Hospital
Other Study IDs: HUS/97/2021
Record Dates: First submitted 2022-01-24; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Post Covid-19 Condition
Keywords: Post Covid-19 condition; long Covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CRP, blood count, sedimentation rate, GT, krea, TSH, fasting glucose, ECG, Alat, Afos, K, Na, Ca, Alb, preAlb, B12-TC, cortisole
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Multiprofessional, tailored rehabilitation — Patients receive individual, tailored, multiprofessional rehabilitation

SUMMARY:
Up to 20% of patients with Covid-19 develop symptoms that last more than 3 months, which is known as long Covid or Post-Covid-19 condition. The mechanism of the long term symptoms is not totally understood although inflammation, autoimmune reactions and thromboembolism are among suspected contributors. At Helsinki University hospital, a long Covid clinic was opened in June 2021. The aim of this cohort study is to monitor the patients that attend the clinic, follow up their functional abilities, quality of life and prognosis.

DETAILED DESCRIPTION:
The patients are asked to give their informed consent for the participation in the cohort study. They fill in a questionnaire before entering the clinic that assesses their symptoms, previous medical history, medications, lifestyle, symptoms, sleep, psychosocial measures including depression, anxiety, resilience and quality of life.

The patients are asked to give blood samples that rule out other diseases that may cause the symptoms. At the clinic, they attend a physician's consultation with physical exam. Later, in another apppointment, a physicotherapist assesses their physicial functioning including 6 minutes walking test and grip strength. They also attend a psychologist who conducts short, 30 min neuro-cognitive testing.

Patients receive psychoeducation of the Post Covid-19 condition and individual, tailored support and rehabilitation. They are given the opportunity to take part in group counselling once a week during 6 weeks.

The patients are followed up by nurse telephone calls at 3, 6 and 12 months as well as by questionnaires via a secured website.

The main outcome measure in this study is functional ability as measured by WHODAS2.0.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosed Covid-19 infection at least 3 mo before entry (either PCR positive or antigen test positive or hospitalisation because of Covid-19)

Exclusion Criteria:

* patients for whom participation would be too exhausting, for example bed patients
* patients who cannot fill in the questionnaires in Finnish

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptoms of long Covid that have lasted at least 3 mo after the primary infection
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of WHODAS2.0 questionnaire as measured at 12 months | 0, 3, 6, and 12 months
  Functional ability measured by WHODAS2.0 which is a measure developed by WHO and has 36 items. The minimum value is 0, the maximum value is 100. Higher score means worse functional ability.

SECONDARY OUTCOMES:
EUROHIS-8 Quality of life | 0, 3, 6, and 12 months
  EUROHIS-8 is an 8-item quality of life measure. The minimum value is 1 and the maximum value is 5. Higher score means better quality of life.
Health related quality of life | 0, 3, 6, and 12 months
  15D is a health related quality of life measure developed in Finland and the main quality indicator of Helsinki University Hospital. Its minimum value is 0 and maximum 1. Higher score means better health related quality of life.
Depression | 0, 3, 6, and 12 months
  PHQ-9 (Patient Health Questionnaire-9) is a 9-item depression scale. The minimum value is 0 and the maximum is 27. Higher score means more severe depression.
Anxiety | 0, 3, 6, and 12 months
  GAD-7 (General Anxiety Disorder-7) measures anxiety. The minimum score is 0 and the maximum score is 30. Higher score means more severe anxiety.
Symptom severity | 0, 3, 6, and 12 months
  PHQ-15 (Patient Health Questionnaire-15) is a somatic symptom subscale that measures somatic symptom (physical) severity. The minimum score is 0 and the maximum score is 30. Higher score means more severe symptom severity.
Resilience | 0, 3, 6, and 12 months
  Resilience Scale 14 measures the five core characteristics of resilience (purpose, perseverance, self-reliance, equanimity, and authenticity). The minimum value is 0 and the maximum value is 100. Higher score means better resilience.
Sleep | 0, 3, 6, and 12 months
  ISI (Insomnia Severity Index) has seven questions. The minimum value is 0 and the maximum value is 28. Higher score means more severe insomnia.
SSD-12, somatic symptom disorder | 0, 3, 6, and 12 months
  SSD-12 (Somatic Symptom Disorder-12) has 12 items. The minimum value 0 and the maximum is 48. Higher score means more severe perceptions related to somatic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Liira, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
We have applied for EU Horizon funding and potentially share data in that project.

REFERENCES:
- [Derived] Virrantaus H, Liira H, Posharina T, Sulg A, Mantyla T, Kanerva M, Laakso S, Sainio M, Malmivaara A, Vuokko A, Varonen M, Venalainen M, Arokoski J. Prognosis of patients with long COVID symptoms: a protocol for a longitudinal cohort study at a primary care referred outpatient clinic in Helsinki, Finland. BMJ Open. 2023 Oct 17;13(10):e072935. doi: 10.1136/bmjopen-2023-072935. PMID 37848295